CLINICAL TRIAL: NCT04273451
Title: A RadioPathomics Integrated Artificial Intelligence System to Predict Tumor Regression Grading of Neoadjuvant Treatment in Locally Advanced Rectal Cancer: A Multicenter, Prospective and Observational Clinical Study
Brief Title: RadioPathomics Artificial Intelligence Model to Predict Tumor Regression Grading in Locally Advanced Rectal Cancer
Acronym: RPAI-TRG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: The Third Affiliated Hospital of Kunming Medical College. (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, wanxiangbo, Associate Professor of Radiation Oncology, Vice Director, Department of Radiation Oncology, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: RPAI-TRG2020
Record Dates: First submitted 2020-02-15; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Rectal Cancer
Keywords: Radiopathomics features; Artificial intelligence; Locally advanced rectal cancer; Tumor regression grading; Neoadjuvant chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, investigators apply a radiopathomics artificial intelligence (AI) supportive model to predict neoadjuvant chemoradiotherapy (nCRT) response before the nCRT is delivered for the patients with locally advanced rectal cancer (LARC). The radiopathomics AI system predicts individual tumor regression grading (TRG) category based on each patient's radiopathomics features extracted from the Magnetic Resonance Imaging (MRI) and biopsy images. The predictive power to classify each patient into particular TRG category will be validated in this multicenter, prospective clinical study.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational clinical study for validation of a radiopathomics integrated artificial intelligence (AI) system. Patients who have been pathologically diagnosed as rectal adenocarcinoma and defined as clinical II-III staging without distant metastasis will be enrolled from the Sixth Affiliated Hospital of Sun Yat-sen University, the Third Affiliated Hospital of Kunming Medical College and Sir Run Run Shaw Hospital Affiliated by Zhejiang University School of Medicine. All participants should follow a standard treatment protocol, including neoadjuvant concurrent chemoradiotherapy (nCRT), total mesorectum excision (TME) surgery and adjuvant chemotherapy. Images of Magnetic Resonance Imaging (MRI) and biopsy hematoxylin & eosin (H&E) stained slides of each patient should be available before nCRT treatment. The tumor region within these images would be delineated manually by experienced radiologists and pathologists. Further, the outlined images will be presented to the radiopathomics AI system to classify each participant into particular tumor regression grading (TRG) category. Here, the American Joint Committee on Cancer and College of American Pathologist (AJCC/CAP) 4-category TRG system is served as the standard. The actual TRG category of each participant will be confirmed based on pathologic assessment after TME surgery. Through comparisons of the predicted TRG and actual TRG category, investigators calculate the prediction accuracy, specificity and sensitivity as well as the F1 score. This study is aimed to develop a reliable and robust AI system to predict pathologic TRG prior to nCRT administration, facilitating response-guided precision therapy for patients with locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed as rectal adenocarcinoma
* defined as clinical II-III staging (≥T3, and/or positive nodal status) without distant metastasis by enhanced Magnetic Resonance Imaging (MRI)
* intending to receive or undergoing neoadjuvant concurrent chemoradiotherapy (5-fluorouracil based chemotherapy, given orally or intravenously; Intensity-Modulated Radiotherapy or Volume-Modulated Radiotherapy delivered at 50 gray (Gy) in gross tumor volume (GTV) and 45 Gy in clinical target volume (CTV) by 25 fractions)
* intending to receive total mesorectum excision (TME) surgery after neoadjuvant therapy (not completed at the enrollment), and adjuvant chemotherapy
* MRI (high-solution T2-weighted imaging, contrast-enhanced T1-weighted imaging, and diffusion-weighted imaging are required) examination is completed before the neoadjuvant chemoradiotherapy
* biopsy H&E stained slides are available and scanned with high resolution before the neoadjuvant chemoradiotherapy

Exclusion Criteria:

* with history of other cancer
* insufficient imaging quality of MRI to delineate tumor volume or obtain measurements (e.g., lack of sequence, motion artifacts)
* insufficient imaging quality of biopsy slides imaging to delineate tumor volume or obtain measurements (e.g., tissue dissection, color anomaly)
* incomplete neoadjuvant chemoradiotherapy
* no surgery after neoadjuvant chemoradiotherapy resulting in lack of pathologic assessment of tumor response
* tumor recurrence or distant metastasis during neoadjuvant chemoradiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population in the study are the patients with LARC, who are intended to receive or undergoing standard, neoadjuvant concurrent chemoradiotherapy with tumor pathologic response unknown.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The prediction accuracy of the radiopathomics artificial intelligence model | baseline
  The prediction accuracy of the radiopathomics artificial intelligence model for classifying each individual into particular AJCC/CAP TRG category will be calculated.

SECONDARY OUTCOMES:
The specificity of the radiopathomics artificial intelligence model | baseline
  The specificity of the radiopathomics artificial intelligence model for classifying each individual into particular AJCC/CAP TRG category will be calculated.
The sensitivity of the radiopathomics artificial intelligence model | baseline
  The sensitivity of the radiopathomics artificial intelligence model for classifying each individual into particular AJCC/CAP TRG category will be calculated.
The F1 score of the radiopathomics artificial intelligence model | baseline
  The F1 score of the radiopathomics artificial intelligence model for classifying each individual into particular AJCC/CAP TRG category will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbo Wan, MD, PhD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University; Xinjuan Fan, MD, PhD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (3):
- China (3):
  - the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Kunming Medical College, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No